CLINICAL TRIAL: NCT01728961
Title: Pharmacology of Artemisinin-Based Antimalarial Therapy Within the Context of Antiretroviral Therapy
Brief Title: Pharmacology of Antimalarial Therapy With or Without Antiretroviral Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow accrual and funding limitations.
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT P1079; U01AI068632 (NIH)
Record Dates: First submitted 2012-09-12; First posted 2012-11-20 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: HIV Infection; Malaria
Keywords: HIV 1; NVP; malaria; Children; Youth; nevirapine; Coartem Dispersible; Artemether; Lumefantrine; Pharmacokinetics
MeSH Terms: conditions — HIV Infections; Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A: AL + NVP -based ARV treatment (Active Comparator): AL given to children who test positive for malaria and are already taking NVP as prescribed by their healthcare provider
  Interventions: Drug: Artemether/Lumefantrine (AL)
- ARM B: AL with No ARV treatment (Active Comparator): AL given to children who do not meet national guidelines for beginning ARV treatment
  Interventions: Drug: Artemether/Lumefantrine (AL)

INTERVENTIONS:
Drug: Artemether/Lumefantrine (AL)
  Other Names: Coartem Dispersible

SUMMARY:
The purpose of this study is to see if taking nevirapine (NVP) for HIV changes the way artemether/lumefantrine (AL) works in children who are co-infected with both HIV and malaria. The brand of AL used in this study is Coartem® Dispersible. This study will compare the blood levels of AL in co-infected children who already take NVP prescribed by their doctor with the co-infected children who do not take anti HIV medicines because they do not meet national guidelines to start them. The study will also assess the safety of using both medications (AL and NVP) in children.

DETAILED DESCRIPTION:
Malaria and HIV are among the two most important global health problems of our time. Malaria accounts for up to 3 million deaths each year, of which 90% occur in Africa where malaria is the leading cause of mortality in young children. Artemisinin-based combination therapy (ACT) are the mainstay of antimalarial therapy throughout much of the world, yet pediatric pharmacokinetic data on the most widely adopted ACT regimen, artemether/lumefantrine (AL) are lacking. Of equal importance is the assessment of key drug-drug interactions in HIV co-infected children as ARVs are known to affect the metabolic enzyme activity responsible for ACT elimination. This study proposes to investigate the drug-drug interaction between the antimalarial artemether/lumefantrine and nevirapine based antiretroviral (ARV) treatment for HIV in children co-infected in resource limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥3 to ≤12 years at entry.
* Documentation of HIV-1 infection defined as positive results from two samples collected at different time points. The same method may be used at both time points. All samples tested must be whole blood, serum or plasma.

Subjects ≤ 18 months of age

The first test may be any of the following:

1. One HIV DNA Polymerase chain reaction (PCR)
2. One HIV RNA (quantitative >5,000 copies/mL or qualitative)
3. One HIV culture (prior to August 2009)
4. One total HIV nucleic acid

If the first test(s) is positive, a second sample collected and tested using any of the tests listed above (except for qualitative RNA assays) in a laboratory participating in an appropriate external quality assurance program and NIH-approved.

Subjects > 18 months of age

The first test may be any of the following:

1. Two rapid antibody tests from different manufacturers or based on different principles and epitopes
2. One rapid antibody test AND one [enzyme immunoassay (EIA) OR Western blot (WB) OR immunofluorescence OR chemiluminescence]
3. One EIA AND one [WB OR immunofluorescence OR chemiluminescence]
4. One HIV DNA PCR
5. One HIV RNA (quantitative >5,000 copies/mL or qualitative)
6. One HIV culture (prior to August 2009)
7. One total HIV nucleic acid

If the first test(s) is positive, a second sample collected and tested using any of the tests listed above (except for qualitative RNA assays) in a laboratory participating in an appropriate external quality assurance program and either CAP/Clinical Laboratory Improvement Amendments (CLIA) approved (for US laboratories) or NIH-approved (for international laboratories).

* Presentation with malaria as indicated by positive smear for malaria parasites along with clinical evidence of infection (fever or history of fever in the past 24 hours) with planned treatment with AL.
* Receiving: (a) NO ARV drugs for at least 4 weeks prior to study entry with no intent to initiate ARVs during the study duration, OR (b) NVP-based combination ARV therapy for at least 4 weeks prior to study entry, with the intent to continue same for duration of the study.
* NOTE: Subjects who are managed with a NVP-based ARV therapy at the time of study enrollment will continue on NVP-based ARV therapy while receiving AL treatment. Children who have NOT met eligibility for ART according to national guidelines (based on known available data at time of enrollment) will be permitted to enroll in the study group of children receiving NO ARV drugs. For this study arm of NO ARV drugs, subjects must not be receiving any ARV drugs currently and they have must not have been on any ARV drugs for at least 4 weeks prior to entry.
* If subject is already on antimalarial medication at time of study entry, no more than 3 doses of either generic AL or brand Coartem® (either standard tablet or the dispersible formulation) may be given prior to study entry. Subjects may have received only the first, second, and/or third dose as a different AL formulation from the study formulation of Coartem® Dispersible. However, the actual dose of artemether and lumefantrine that has been administered MUST be the same as that stipulated by the protocol.
* Female subjects of reproductive potential (having reached menses, or not having reached menopause or not having undergone hysterectomy, bilateral oophorectomy, or tubal ligation) who engage in sexual activity that could lead to pregnancy must agree to avoid pregnancy during the entire 42 day trial and to consistently and appropriately use at least two of the following contraception methods: condoms, diaphragm or cervical cap with spermicide, intrauterine device (IUD), hormonal-based contraception. A list of acceptable methods can be found in the FDA Birth Control Guide accessible at: http://www.fda.gov/womens
* Note: "Female subjects of reproductive potential" is defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months (e.g. who have had menses within the preceding 24 months), or have not undergone a sterilization procedure (hysterectomy, bilateral oophorectomy or salpingotomy). If the female subject is not of reproductive potential, she is eligible without requiring contraception.
* Demonstrated ability and willingness to swallow study medications.
* Parent or legal guardian able and willing to provide signed informed consent.
* Ability and willingness to complete study procedures and follow-up at the same study site.

Exclusion Criteria:

* Subjects with ≥ Grade 3 hemoglobin abnormalities (toxicities will be graded by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, dated December 2004, Clarification August 2009, must be used and is available on the Regulatory Support Center (RSC) web site (http://rsc.tech-res.com/safetyandpharmacovigilance/).
* Severe malnutrition will be defined as (i) body mass index (BMI) Z-score< -3 Standard Deviations for children ≥5 years old or (ii) Weight-for-Height <-3 Standard Deviations for children <5 years old. (See Appendix IV).
* Note: Children will be evaluated for malnutrition at the time they present for study enrollment when screening evaluations are performed.
* Receipt of a protease inhibitor or efavirenz (EFV) within 4 weeks prior to study entry.
* Subjects not on ART, but who qualify for ART, according to national guidelines (based on all data available at time of enrollment).
* Use of AL for prior episode of malaria within 6 weeks of study entry.
* Currently receiving an antimalarial drug other than AL.
* Pregnancy or breastfeeding
* Signs or evidence of severe malaria. Severe malaria is defined as:

  * Unarousable coma (if after convulsion, > 30 minutes)
  * OR ANY TWO OF THE FOLLOWING SYMPTOMS:
  * Recent febrile convulsions (within 24 hours)
  * Altered consciousness (confusion, delirium, psychosis, coma)
  * Lethargy
  * Unable to drink
  * Unable to stand/sit due to weakness
  * Severe anemia (Hb < 5.0 gm/dL)
  * Respiratory distress (labored breathing at rest)
  * Jaundice
* Repeated vomiting that, in the opinion of the investigator, would interfere with oral administration and drug absorption.
* Current treatment for malignancy.
* Known allergy or intolerance to milk products
* In the case where a seemingly eligible participant who is small, has a known or planned blood draw, or will have blood drawn for any reason, such that the total volume blood being drawn over any 8 week period will exceed 9.5 mL/kg. (See Appendix II).
* Any disallowed medications (see Section 4.3) used within 3 weeks of study entry.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time zero to last quantifiable concentration (AUC) | NVP PK: At study entry and study day 3, AL PK: At study days 3, 4, 8, and 14
  Area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration
Toxicity | At study entry and study days 28 and 42
  Number of subjects with adverse events of Grade 3 or higher will be recorded
Maximum observed plasma concentration (Cmax) | NVP PK: At study entry and study day 3, AL PK: At study days 3, 4, 8, and 14
  Maximum observed plasma concentration computed for each individual and then summarized for the strata
Minimum observed plasma concentration (Cmin) | NVP PK: At study entry and study day 3, AL PK: At study days 3, 4, 8, and 14
  Minimum observed plasma concentration computed for each individual and then summarized for the strata
Toxicity | At study days 28 and 42
  Percentage of subjects with adverse events of Grade 3 or higher will be recorded Safety Issue: Yes

SECONDARY OUTCOMES:
HIV-1 Viral Load | At study entry and study days 8, 14, and 42
  Dried Blood Spot (DBS) samples will be collected on all study subjects for HIV-1 viral load measurement.
NVP resistance | At study entry and study day 42
  Dried Blood Spot (DBS) samples will be collected on all subjects. Drug resistance testing will only be performed on subjects who show changes in viral load pattern between study entry and study day 42.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Aweeka, Pharm.D., Principal Investigator — IMPAACT/UCSF
Locations (3):
- Malawi (2):
  - College of Med. JHU CRS (30301), Blantyre, Blantyre
  - University of North Carolina Lilongwe (12001), Lilongwe
- Makerere University - JHU Research Collaboration (30293), Kampala, Uganda